CLINICAL TRIAL: NCT06821412
Title: Wireless Non-Invasive Advanced Control of Microprocessor Prostheses and Orthoses II
Brief Title: Wireless Prosthetic Control Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: University of Hartford (Other); Worcestor Polytechnic Institute (WPI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: IRB-23-0722; W81XWH22C0049 (Other Grant/Funding Number: U.S. Army Medical Research Acqisition Activity (USAMRAA))
Record Dates: First submitted 2025-01-17; First posted 2025-02-12 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Prostheses; Upper Limb Amputation Below Elbow

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wireless Control (Experimental): The participant wears the experimental socket in the wireless configuration using the prototype ASTERISK system connected within the electronics of the prosthetic socket. The electronics are not accessible by the participant which allows both configurations to be blinded to the participants.
  Interventions: Device: ASTERISK System
- Wired Control (Sham Comparator): The participant wears the experimental socket in the wired configuration, which mimics the current setup for EMG-controlled prostheses. The electronics are not accessible by the participant which allows both configurations to be blinded to the participants.
  Interventions: Device: Wired Configuration

INTERVENTIONS:
Device: ASTERISK System — This intervention uses an experimental socket fabricated by a certified prosthetist. The electronics within the experimental socket are set up with the ASTERISK system, which sends information collected from the EMG sensors to the prosthetic hand wirelessly rather than the current available method of wired control.
  Arms: Wireless Control
Device: Wired Configuration — This intervention uses the same experimental socket that is used for the ASTERISK intervention. The prosthesis is set-up with wired EMG control, which is the current available method for EMG-controlled prostheses.
  Arms: Wired Control

SUMMARY:
The goal of this proposed project is to evaluate the effectiveness of our novel wireless electrode system, which the investigators refer to as the Asterisk system, on transradial prosthesis users. There are numerous benefits to the upper limb prosthesis community being able to utilize wireless electrodes. These benefits include allowing for the use of a prosthetics liner to assist with fit and comfort, easier implementation of electromyography (EMG) controlled (also referred to as myoelectric control) prosthesis for individuals with osseointegration, and additional EMG electrode location options if the muscle activity captured within the prosthetic socket does not provide reliable prosthesis control. The investigators intend to use this data to develop the Asterisk wireless electrode system into a commercial product. The findings will also be shared with the research community to help drive the design of future devices.

DETAILED DESCRIPTION:
The study evaluates the Asterisk system to determine if Asterisk will increase a user's self-reported satisfaction with their prosthesis as measured by the Orthotic and Prosthetic User Survey-Satisfaction with Device (OPUS-SD) when compared to their current prosthesis. While the technology has the potential to benefit other patient populations, the investigators will focus this initial pilot study on individuals with trans-radial limb absence to reduce potential confounding variables associated with including other amputation levels.

The proposed Asterisk system would allow for liners to be worn with upper limb myoelectric systems. By creating wireless sensors that can be worn under a liner, the sensors can be placed on the skin to collect the myoelectric signal, the liner then rolled over the top of the sensors when donning, and the sensors can transmit the EMG signal wirelessly to the prosthesis. The Asterisk system would also be beneficial to those with osseointegration, unreliable prosthesis control with EMG signals collected in the area encompassed by their socket, and prosthesis users who struggle with volume management.

The investigators plan to conduct a randomized 2x2 crossover study to evaluate benefits provided by prostheses utilizing the Asterisk electrodes over standard prostheses. The two crossover test conditions are "Experimental" (myoelectric control with the Asterisk system) and "Control" (standard prosthetic device configuration). For the control condition, the subject will be using their everyday prosthesis. For the experimental condition, the investigators will fabricate and provide a new socket to allow for the additional socket volume necessary for liners worn with the Asterisk electrodes. Each subject will participate in both conditions of the study. The condition that each subject completes first will be chosen by a random number generator that also ensures block randomization with an equal number of participants assigned to each condition first in the test sequence using a custom program that was created under a prior research project.

Subjects will participate in at least four research visits and will take part in two, one-month long take-home periods. Some researchers have suggested that persons with transradial amputation require, on average, 3-5 weeks of training , while others have suggested that 5 hours of training is sufficient . Therefore, the investigators expect a one-month take-home period to be sufficient to allow users to become comfortable with each socket configuration while optimizing the take-home duration to maximize study efficiency.

In-lab test visits will consist of outcome measures such as the OPUS-SD and the Box and Blocks functional test for each study condition.

After receiving IRB approval, subjects will be recruited and screened for eligibility. If they are eligible and decide to participate, they will be scheduled for their first site visit. At the first study visit, subjects will be given the informed consent form to read through entirely before signing and are encouraged to ask questions at any time.

All subjects, regardless of test condition, will then receive training on controlling their prosthesis in their current test condition by the study personnel. The training will start with basic skills, including opening and closing the device, and grasping various shapes such as cone/cups, regular/irregular block shapes, and various size and weight balls. Then they will advance to splinter skills, involving partial completion of activities of daily living (ADL) tasks, for example, positioning the device on the handle of a large mug and gripping the handle. And finally, they will practice full task skills, e.g., grasping the handle of a large mug and bringing the mug up to the subject's mouth to drink from it, putting the mug back down, and releasing the grip. All subjects will also receive instructions on how to fill out the daily log (for the ensuing at-home portion of the study).

In certain cases, subjects may become too fatigued (physically or mentally) to complete the entire planned activity during the scheduled visit. Additionally, in some cases, equipment failures may delay completion of the activity planned for a visit. In such a case, subjects may be invited to return to complete the visit activity at the next mutually agreed date. If the return visit is due to equipment failures, subjects will be offered the standard travel stipend for the secondary visit.

During take-home periods, the investigators will periodically check-in with the subject (by phone, text, email, etc.) to maximize adherence to the daily log, debug any technical issues, etc.

ELIGIBILITY:
Inclusion Criteria:

* current wearers of trans-radial myoelectric prostheses or orthoses
* have used their prostheses/orthoses for at least six months
* understand spoken and written English (for the purpose of consenting)

Exclusion Criteria:

* have any neurological or physical conditions which would prevent them from performing the experimental tasks
* are pregnant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin McDonald, Principal Investigator — Liberating Technologies, Inc.
Locations (1):
- Liberating Technologies, Inc., Holliston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Wireless Control, Then Wired Control: The participant wears the experimental socket in the wireless configuration using the prototype ASTERISK system connected within the electronics of the prosthetic socket. Then the participant wears the experimental socket in the wired configuration, which mimics the current setup for EMG-controlled prostheses The electronics are not accessible by the participant which allows both configurations to be blinded to the participants.
  ASTERISK System: This intervention uses an experimental socket fabricated by a certified prosthetist. The electronics within the experimental socket are set up with the ASTERISK system, which sends information collected from the EMG sensors to the prosthetic hand wirelessly rather than the current available method of wired control.
  Wired Configuration: This intervention uses the same experimental socket that is used for the ASTERISK intervention. The prosthesis is set-up with wired EMG control, which is the current available method for EMG-controlled prostheses.
- Wired Control, Then Wireless Control: The participant wears the experimental socket in the wired configuration, which mimics the current setup for EMG-controlled prostheses. Then the participant wears the experimental socket in the wireless configuration using the prototype ASTERISK system connected within the electronics of the prosthetic socket. The electronics are not accessible by the participant which allows both configurations to be blinded to the participants.
  ASTERISK System: This intervention uses an experimental socket fabricated by a certified prosthetist. The electronics within the experimental socket are set up with the ASTERISK system, which sends information collected from the EMG sensors to the prosthetic hand wirelessly rather than the current available method of wired control.
  Wired Configuration: This intervention uses the same experimental socket that is used for the ASTERISK intervention. The prosthesis is set-up with wired EMG control, which is the current available method for EMG-controlled prostheses.
Period: Overall Study
Arm/Group | Wireless Control, Then Wired Control | Wired Control, Then Wireless Control
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wireless Control, Then Wired Control | Wired Control, Then Wireless Control | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Orthotics and Prosthetics User Survey - Satisfaction With Device (OPUS-SD)
Description: The Orthotics and Prosthetics User's Survey (OPUS) is a self-report questionnaire consisting of five modules. The version of the OPUS which will be administered consists of 9 questions in 1 category (satisfaction with device). Questions are asked and scored on a scale from 0-4 (0=strongly disagree, 1=disagree, 2=neither agree nor disagree, 3=agree, and 4=strongly agree), with a higher value indicating a better outcome. There is an additional response for "Don't know / Not Applicable", which if chosen, is not included in the scoring.
  This survey will be given at the end of each study condition (2 conditions, 1 month per condition).
  Analysis is reported as a value that calculates the average of all questions (sum up all questions and divide by total number of questions).
Time Frame: At the end of each 1 month condition
Population: 4 total participants enrolled, 4 total completed each condition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wireless Control | Wired Control
Number analyzed (Participants) | 4 | 4
score on a scale | 2.89 (0.94) | 3.11 (0.77)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/collected during each condition. With each condition lasting about 1 month, each participant was monitored for adverse events for about 3 months total. Adverse events were monitored/assessed as needed, with study staff checking in more frequently if participants reached out with questions. Participants were told to reach out to study staff immediately if adverse events did occur.
Arm/Group | Wireless Control | Wired Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT06821412/Prot_SAP_000.pdf